CLINICAL TRIAL: NCT04496609
Title: Assessment of the Efficacy and Safety of Epidural Electrical Stimulation of the Lumbosacral Spinal Cord in the Symptomatic Treatment of Motor, Vesico-sphincter and Genito-sexual Disorders in Patients With Incomplete Spinal Cord Injuries
Brief Title: Assessment of the Efficacy and Safety of EESS in Patients With Incomplete Spinal Cord Injuries
Acronym: Parastim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016/50
Record Dates: First submitted 2020-07-20; First posted 2020-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation-automated rehabilitation/automated rehabilitation (Experimental): * Stimulation and automated rehabilitation (2 sessions of 45 minutes per day) for 40 working days
  * Washout 30 days
  * Automated rehabilitation (2 sessions of 45 minutes per day) for 40 working days
  Interventions: Device: Stimulation and automated rehabilitation / automated rehabilitation
- Automated rehabilitation/Stimulation-automated rehabilitation (Experimental): * Automated rehabilitation (2 sessions of 45 minutes per day) for 40 working days
  * Washout 30 days
  * Stimulation and automated rehabilitation (2 sessions of 45 minutes per day) for 40 working days
  Interventions: Device: Automated rehabilitation / Stimulation and automated rehabilitation

INTERVENTIONS:
Device: Stimulation and automated rehabilitation / automated rehabilitation — Stimulation and automated rehabilitation for 40 working days, then washout during 30 days, then automated rehabilitation for 40 working days
  Arms: Stimulation-automated rehabilitation/automated rehabilitation
Device: Automated rehabilitation / Stimulation and automated rehabilitation — Automated rehabilitation for 40 working days, then washout during 30 days, then automated rehabilitation for 40 working days
  Arms: Automated rehabilitation/Stimulation-automated rehabilitation

SUMMARY:
Neurological disability caused by traumatic lesions of the spinal cord is a significant challenge for medicine and society. These lesions, leading to sublesional central nervous system dysfunction, include sensorimotor, vesico-sphincter and genito-sexual disorders. To date, there is no treatment that enables spinal cord function to be restored.

Preclinical studies have been able to demonstrate the recovery of locomotor activity with a combination of locomotor training, pharmacological intervention and epidural electrical stimulation of the lumbosacral spinal cord (EESS) in adult rats with spinal cord transection. An American team have recently been able to show that EESS, combined with locomotor training, caused neurological improvement in four paraplegic patients, with electromyographic muscular activation patterns similar to those observed during walking. In fact, these authors also showed an improvement, under stimulation, of the VS and GS functions, but with no detailed documentation.

Starting with a conceptual and preclinical rationale, and with proof of clinical concept demonstrated in several reported cases, we propose a clinical trial with an original cross-over design to validate the hypothesis that EESS combined with training in patients with incomplete spinal cord injuries would, with a good tolerance profile, allow motor, vesico-sphincter (VS) and genito-sexual (GS) disorders to be restored in patients with incomplete spinal cord injuries.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years inclusive
* Male or female
* Incomplete ASIA B or C spinal cord lesion with level of lesion located above T10 (sensation preserved below level of lesion)
* Absence of significant motor deficit of the upper limbs or recovered motor deficit (muscular score ≥ 4/5)
* Patient with spinal cord injury at least 2 years old and considered stable not walking
* Spinal cord lesion determined by spinal cord MRI (intramedullary hypersignal)
* Patient who can benefit from an iterative rehabilitation programme
* Patient with stable health condition with no cardiopulmonary disease
* Patient with orthopaedic condition compatible with verticality and walking
* Persistence of adductor reflexes up to L2
* Patient with no current neuromodulation implant: spinal cord neurostimulator, brain, peripheral nerve or intrathecal treatment
* Patient with no coagulopathy, cardiac risk factors or other medical risk factors significant for surgery
* Local anatomical conditions compatible with implantation of the epidural electrode (determined by MRI of the spinal cord)
* Person who benefits from or is entitled to a social security scheme
* Having provided signed informed consent

Exclusion Criteria:

* Significant cerebral lesion on a previous cerebral MRI
* Psychiatric or cognitive disorder history (known or detected during the consultation with the psychologist)
* Protected adult patients
* Pregnant (determined by a negative pregnancy test) or breastfeeding women
* Respiratory failure (vital capacity < 50%) (surgery in prone position)
* Repeated urinary infections (≥3 per year)
* Planned absence that may hinder participation in the study (travelling abroad, relocation, imminent moving)
* Patients with spasms (PENN scale > 2)
* Cauda equina syndrome
* Patients presenting with a contraindication to an MRI being carried out: i) pacemaker, ii) non-MRI-compatible heart valve, iii) clips, stents, coils, etc. that are not MRI-compatible, iv) cochlear implant, v) metal foreign body, etc.)
* Patients presenting with a contraindication to MEPs being carried out (notably wearing of ferromagnetic material, heart stimulator)
* Patients on oral anticoagulants
* Patients with botulinic toxin injection
* Patients with bedsore
* Undernourished patients (BMI < 19)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of number of patients able to move over a distance of 5 metres | through study completion
  Determined by a capability to move over a distance of 5 metres with or without technical aid, with the option of stopping on the way

SECONDARY OUTCOMES:
Percentage of patients capable of moving at the end of treatment | 1 hour
  Based on the rehabilitation programme over a distance of 5 metres with or without technical aid, with the option of stopping on the way, Surface EMG, Bipodal balance measurement
Assessment of vesico-sphincter function | 1 hour
  Measurement using cystomanometry, flow measurement and assessment of post-micturition residue by means of a bladder scan
Assessment of the genito-sexual function | 30 minutes
  Measurement with MSHQ (Male Sexual Health Questionnaire) scale in men and FSFI (Female Sexual Function Index) in women MSHQ scale: minimum value (worse outcome): 7 - maximum value (better outcome): 80 FSFI scale: minimum value:2 (worse outcome) - maximum value: 36 (better outcome)
Assessment of the excitability of the spinal neuronal circuits | 1 hour
  Measurement of the reciprocal inhibition directed from the tibialis anterior to the soleus and the presynaptic inhibition applied to the fibres of the soleus by modifying the range of the soleus H-reflex obtained by percutaneous peripheral nerve electrical stimulation
Assessment of the kinetics of action of the induced effects | 1 hour
  Assessment according to the epidural electrical stimulation paradigms
Assessment of capability to move over a distance of 5 metres at the end of washout period for treatment combining EESS and rehabilitation program | throughout the study
  Measurement of covered distance at the end of washout period for treatment combining EESS and rehabilitation program
Assessment of capability to move over a distance of 5 metres at the end of washout period for rehabilitation program | 30 minutes
  Measurement of covered distance at the end of washout period for rehabilitation program
Assessment of capability to move over a distance of 5 metres after 6 months of treatment | Month 6
  Measurement of covered distance after 6 months of treatment
Assessment of vesico-sphincter function at the end of washout period for treatment combining EESS and rehabilitation program | 1 hour
  Measurement using cystomanometry, flow measurement and assessment of post-micturition residue by means of a bladder scan
Assessment of vesico-sphincter function at the end of washout period for rehabilitation program | 1 hour
  Measurement using cystomanometry, flow measurement and assessment of post-micturition residue by means of a bladder scan
Assessment of vesico-sphincter function after 6 months of treatment | Month 6
  Measurement using cystomanometry, flow measurement and assessment of post-micturition residue by means of a bladder scan
Assessment of the genito-sexual function at the end of washout period for treatment combining EESS and rehabilitation program | 30 minutes
  Measurement with MSHQ (Male Sexual Health Questionnaire) scale in men and FSFI (Female Sexual Function Index) in women MSHQ scale: minimum value (worse outcome): 7 - maximum value (better outcome): 80 FSFI scale: minimum value:2 (worse outcome) - maximum value: 36 (better outcome)
Assessment of the genito-sexual function at the end of washout period for rehabilitation program | 30 minutes
  Measurement with MSHQ (Male Sexual Health Questionnaire) scale in men and FSFI (Female Sexual Function Index) in women MSHQ scale: minimum value (worse outcome): 7 - maximum value (better outcome): 80 FSFI scale: minimum value:2 (worse outcome) - maximum value: 36 (better outcome)
Assessment of the genito-sexual function after 6 months of treatment | Month 6
  Measurement with MSHQ (Male Sexual Health Questionnaire) scale in men and FSFI (Female Sexual Function Index) in women MSHQ scale: minimum value (worse outcome): 7 - maximum value (better outcome): 80 FSFI scale: minimum value:2 (worse outcome) - maximum value: 36 (better outcome)
Assessment of the excitability of the spinal neuronal circuits at the end of washout period for treatment combining EESS and rehabilitation program | 1 hour
  Measurement of the reciprocal inhibition directed from the tibialis anterior to the soleus and the presynaptic inhibition applied to the fibres of the soleus by modifying the range of the soleus H-reflex obtained by percutaneous peripheral nerve electrical stimulation
Assessment of the excitability of the spinal neuronal circuits at the end of washout period for rehabilitation program | 1 hour
  Measurement of the reciprocal inhibition directed from the tibialis anterior to the soleus and the presynaptic inhibition applied to the fibres of the soleus by modifying the range of the soleus H-reflex obtained by percutaneous peripheral nerve electrical stimulation
Assessment of the excitability of the spinal neuronal circuits after 6 months of treatment | 1 hour
  Measurement of the reciprocal inhibition directed from the tibialis anterior to the soleus and the presynaptic inhibition applied to the fibres of the soleus by modifying the range of the soleus H-reflex obtained by percutaneous peripheral nerve electrical stimulation
Assessment of quality of life | 30 minutes
  Measurement with EQ5D-3L (EuroQol 5 Dimensions - 3 Levels) scale
Number of patient with AE/SAE related to tolerance | through study completion
  Reporting of AE and SAE
Number of patient with AE/SAE related to safety | through study completion
  Reporting of AE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: Béchir Jarraya, MD, Principal Investigator — Hôpital Foch
Locations (2):
- France (2):
  - Hôpital Raymond Poincaré, Garches
  - Hôpital Foch, Suresnes